CLINICAL TRIAL: NCT01488136
Title: Use of Diazoxide in Acute Hypoglycaemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2010DM03; 2011-005011-93 (EudraCT Number)
Record Dates: First submitted 2011-10-26; First posted 2011-12-08 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Hypoglycaemia; Diazoxide
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Diazoxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diazoxide (Active Comparator): Oral diazoxide 7 mg/kg
  Interventions: Drug: Diazoxide
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diazoxide — Diazoxide 7mg/kg, given 2 hours before the start of the clamp study
  Other Names: Eudemine (Diazoxide)
  Arms: Diazoxide
Drug: Placebo — Lactose Ph capsules (Placebo)
  Other Names: Lactose Ph capsules (Placebo)
  Arms: Placebo

SUMMARY:
The investigators know that intensive insulin therapy and tight glucose control is associated with reduction of diabetic complications. However, many patients on insulin don't achieve this because of the risk and the fear of hypoglycaemia (too low blood glucose).

There has been a lot of work done recently looking at the mechanisms by which the brain detects hypoglycaemia. A key player is a potassium channel in the brain (KATP channel). Studies have shown that when these channels are opened, there is a release of hormones such as adrenaline that can help in raising blood sugars to counteract and increase awareness of hypoglycaemia. The investigators study aims to look at an old drug called diazoxide, which is able to open KATP channels.

The investigators aim to see if diazoxide will amplify the release of hormones such as adrenaline when the blood sugar is low. If this is the case, this will aid quicker recovery following hypoglycaemia.

The investigators aim to do this by performing a well established experimental protocol that has been performed safely over the last 20 years called a clamp study. The clamp study will involve slowly bringing the blood sugars down using insulin and intravenous glucose in a controlled fashion. The main outcome will be the hormonal responses (adrenaline response) at a blood sugar level of 2.5mmol/L. Symptoms of hypoglycaemia will be monitored, as well as working memory tests using standardised questionnaires.

The design of the investigators study will be a randomised trial comparing the effects of diazoxide with placebo in which all patients will receive both diazoxide and placebo in random order (crossover design).

DETAILED DESCRIPTION:
This will be conducted in a double blinded (neither subject nor the researcher will know the order of the IMP(drug/placebo). All subjects will receive both the active drug and placebo in a random fashion (crossover design).

Once identified, patients will be given a participant information sheet. They will be contacted at a later date (minimum 24 hours) to determine if they are willing to participate in the trial.

Subjects will then be consented, and attend a screening visit, where it will be ascertained whether they fit the inclusion/exclusion criteria. Further details of the study will also be given to them at this visit. They will then attend a few days before the first study, and will be shown how to use the continuous glucose monitor which will measure their glucose overnight, prior to the start of the study. The reason for this, is that if they have very low blood sugars the night before the study, this can influence the results of the study, and they will be given an alternative day to attend. Provided they have been free of any hypoglycaemic episodes, the night before, they can then proceed with the study.

On the day of the study,we will place two intravenous cannulae. The cannulae in the hand vein will be placed in a warm chamber, in order to make it more more reflective of sampling at the blood brain barrier.

The subject will either have the investigational medicinal product (diazoxide) or placebo. Blood pressure and heart rate will be monitored throughout the clamp study. After 2 hours, with the use of insulin and dextrose, the subject's blood sugar will be brought to near normal and kept there for 40 minutes. After this, the blood sugar will be dropped in stages, until a blood sugar of 2.5mmol/L is reached. The blood sugar will be monitored very closely, with 5 minute sampling taken through one of the cannulue in situ, to avoid repeated stabbing. Also at regular intervals, blood samples will be taken for measurement of hormones, including adrenaline. At each stage, subjects will be asked about symptoms they are experiencing and a series of verbal working memory tests will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (aged 18-55) with >5 years disease duration
* On intensive insulin therapy (CSII or multiple daily injections)
* HbA1C<8.0%
* Ability to give written informed consent to participate in the study
* BMI between 20-29

Exclusion Criteria:

* History of significant cardiac, hepatic, renal or neurological disease.
* Significant head injury, epilepsy or hypoglycaemia-induced seizures.
* Pregnancy.
* Breast feeding mothers.
* Participants on thiazide diuretics
* Participants on other potassium channel openers (nicorandil, minoxidil)
* Participants on medications with vasodilatory properties such as methyldopa, reserpine, theophyllines and nitrites.
* Participants on hydantoins (fosphenytoin, phenytoin)
* Significant anaemia Hb<11.0 and Hct<33%.
* If they have donated blood in the last 30 days.
* All those who have participated in a CTIMP in the last 3 months
* Participants who are already on diazoxide or who have a past history of allergy to diazoxide

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Adrenaline response(pmol/L) at 2.5mmol/L of glucose | 1 year
  The body secretes hormones such as adrenaline as a response to low blood sugars. Patients who have had insulin-dependant diabetes for over 5 years rely heavily on adrenaline release, to produce symptoms, so that they can respond appropriately to low blood sugars. However, this response is blunted in those with type 1 diabetes.
  Our question is whether the magnitude of this response can be increased by use of diazoxide in the context of hypoglycaemia, so that patients with insulin-dependant diabetes become better aware of hypoglycaemia.

SECONDARY OUTCOMES:
Glucose Thresholds (calculated when counter-regulatory hormone release is greater than 2SD of hormone level at euglycaemia 4.0mmol/L blood sugar) of each of the counter-regulatory hormones (adrenaline, noradrenalin, glucagon) | 1 year
  Our study design enables us to bring down the blood sugar in a controlled fashion and maintain it at certain levels. We will be measuring hormones including adrenaline and testing cognitive function as well as assessing symptoms at each of these blood sugar levels. We want to see if diazoxide affects the threshold at which patients are able to mount a clinically relevant rise in counter-regulatory hormones and symptoms of hypoglycaemia.

OTHER OUTCOMES:
Symptom scores and Cognitive function scores at 2.5mmol/L | Done during the hyperinsulinaemic hypoglycaemic clamp
  Symptom scores will be assessed using the Edinburgh Hypoglycaemia Symptom score assesment, and Cognition will be assessed using Trail Making B, Digit substituition, Digit forward and backward and 4 choice reaction tests.

CONTACTS AND LOCATIONS:
Overall Officials: Rory J McCrimmon, MD, Study Chair — Clinical Reader; Priya S George, MRCP, Principal Investigator — Clinical Research Fellow
Locations (1):
- NHS Tayside, Dundee, United Kingdom

REFERENCES:
- [Background] George PS, Tavendale R, Palmer CN, McCrimmon RJ. Diazoxide improves hormonal counterregulatory responses to acute hypoglycemia in long-standing type 1 diabetes. Diabetes. 2015 Jun;64(6):2234-41. doi: 10.2337/db14-1539. Epub 2015 Jan 15. PMID 25591873